CLINICAL TRIAL: NCT03938532
Title: Feasibility and Impact of Volume Targeted Ventilation for Preterm Infants Born <32 Weeks Gestational Age With Need for Invasive Positive Pressure Ventilation in the Delivery Room in Reducing Neonatal Pulmonary Morbidities
Brief Title: Feasibility and Impact of Volume Targeted Ventilation in the Delivery Room
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinuation of the study Product by manufacturer
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Ruben, Associate Professor of Pediatrics, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BH-19-006
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Prematurity; BPD - Bronchopulmonary Dysplasia; Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: 2 parallel arm
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control Arm (Active Comparator): Infant will receive pressure regulated breaths, 40-60 breaths/min, PiP of 20-24cm of water as recommended by 2017 Neonatal Resuscitation Program (NRP) guidelines. Reading of the TV will be blinded from the providers as in routine clinical situations
  Interventions: Device: Tidal Volume Measurement using the Philips Respironics NM3 monitor
- Intervention Arm (Experimental): Infants in the intervention arm will receive VTV following intubation. Peak inspiratory pressure (PiP) provided via T-piece resuscitator will be visible to the providers, and the provider can regulate the PiP to achieve the desired TV goal (4-6 ml/kg), at a rate of 40-60 breaths/min
  Interventions: Device: Volume Targeted Ventilation (VTV) using the Philips Respironics NM3 monitor

INTERVENTIONS:
Device: Volume Targeted Ventilation (VTV) using the Philips Respironics NM3 monitor — Infants in the intervention arm will receive VTV following intubation. Peak inspiratory pressure (PiP) provided via T-piece resuscitator will be visible to the providers, and the provider can regulate the PiP to achieve the desired TV goal (4-6 ml/kg), at a rate of 40-60 breaths/min
  Arms: Intervention Arm
Device: Tidal Volume Measurement using the Philips Respironics NM3 monitor — Tidal Volume Measurement using the Philips Respironics NM3 monitor
  Arms: Control Arm

SUMMARY:
Despite significant improvement in preterm infant survival, the incidence of bronchopulmonary dysplasia (BPD) in infants born < 28 weeks gestational age (GA) has been relatively stable at ~40%, with 10,000-15,000 new cases estimated annually. Delivery room (DR) management of preterm infants during the initial resuscitation has a significant impact on future development of BPD. Current DR practice as recommended by the Neonatal Resuscitation Program (NRP), focuses on providing positive pressure ventilation (PPV) for intubated infants based on pressure limited ventilation (PLV). But with rapidly changing pulmonary compliance during the early newborn period, PLV may lead to under or over inflation of the lungs and induce significant volutrauma, barotrauma and/or atelectotrauma, all of which are associated in the pathogenesis of BPD. No studies have specifically reported tidal volume (TV) provided in the DR in intubated infants with current PLV practices. Similarly, no study has evaluated the safety and efficacy of volume targeted ventilation (VTV) in the DR and its impact on BPD.

With the proposed study, in Phase I, the investigators aim to demonstrate that measuring TV in intubated infants receiving PPV via PLV is feasible. The investigators also seek to demonstrate that with PLV, TV is highly variable in the first few hours of life, even with the same peak inspiratory pressures (PiP) due to rapidly changing pulmonary compliance. A successful Phase I will demonstrate that measuring TV is feasible in the DR, and with information on real time actual TV achieved during PPV, it is possible to target the TV for a goal TV by adjusting the PiP provided.

Phase II will be a pilot randomized control trial to demonstrate feasibility of VTV compared to PLV. The investigators will also aim to understand the pulmonary mechanics and physiology during VTV. A successful Phase II will demonstrate VTV is feasible, is associated with stable TV, decreased peak inspiratory pressure and oxygen needs compared to PLV, and not associated with increased complications compared to PLV. It will thereby justify a larger randomized control trial with enough power to evaluate the efficacy of VTV in reducing BPD and other long term pulmonary morbidities for preterm infants.

DETAILED DESCRIPTION:
BACKGROUND BPD continues to be one of the most common complications associated with preterm birth. A 2013 US study reported an increase in healthcare cost of $31,565 associated with BPD, after controlling for birth weight, gestational age, and socio-demographic characteristics during the initial neonatal intensive care unit (NICU) hospitalization itself. This economic burden starts from the initial NICU admission and persists through childhood and adulthood. A recent Spanish study published in 2013, reported that the healthcare related cost during the first 2 years of life of a preterm baby with BPD and no other major prematurity-related complications ranged between €45,049.81 and €118,760.43, in Spain, depending on birth weight and gestational age. If the baby required home oxygen therapy or developed pulmonary hypertension, this cost could further escalate to €181,742.43. With 10,000-15,000 new cases of BPD annually in USA alone, the economic impact of BPD is tremendous.

The pathogenesis of BPD is multifactorial, with lung injury from mechanical ventilation, oxygen toxicity, and antenatal or postnatal infections, all leading to lung inflammation which play a key role in the development of BPD. Delivery room (DR) management of preterm infants during the initial resuscitation is critical, and can have a significant impact on development of BPD. Studies have demonstrated that DR respiratory management with invasive respiratory support and higher oxygen content is associated with increased risk of death and/or BPD compared to non-invasive ventilation and lower oxygen resuscitation, respectively. Preterm infants stabilized on continuous positive airway pressure (CPAP) with prudent titration of supplemental oxygen in the delivery room to achieve targeted oxygen saturations have demonstrated improved rates of BPD.

CURRENT STANDARD OF PRACTICE Current DR practice for intubated preterm infants focuses on pressure limited ventilation using either a self-inflating bag or a T-piece resuscitator where the provider regulates the inflation pressure and inflation time, but not the tidal volume.

As an infant transitions to extra uterine life, pulmonary compliance changes rapidly. Total pulmonary compliance is a composite of the lung and chest wall compliances. In preterm infants, the chest wall is composed primarily of cartilage rendering the chest wall highly compliant, and as a result, the neonatal lung is more prone to collapse. Preterm lungs additionally have reduced surfactant production which further decreases lung compliance. Upon initiation of positive pressure ventilation (PPV), the rapid fluid shift in the immediate newborn period can also result in swift changes in a newborn's pulmonary compliance. Provision of maternal antenatal steroids as well as surfactant replacement therapies can positively impact the preterm pulmonary outcomes. For these preterm infants, tidal volumes generated during PPV is directly proportional to the lung compliance as demonstrated by the formula: Cdyn=VT/(PiP-PEEP), where, VT = tidal volume; PIP=peak inspiratory pressure; and PEEP=positive end-expiratory pressure.

Hence, with PLV the exact same pressure due to rapidly changing lung compliance may lead to under-inflation or over-inflation of the lungs.

Once admitted in the NICU, providing VTV to preterm infants is standard practice in the investigators NICU, with inter-provider preference over volume versus pressure ventilation, with no true consensus. However, in the DR the practice continues to be utilizing PLV and with the proposed study, the investigators seek to provide physiologically more appropriate VTV to the preterm infants right from the birth in the DR.

SIGNIFICANCE With rapidly changing lung compliance in the immediate neonatal transition phase, PLV can lead to significant variability in the delivered TV. Recent reports suggests that pressure limited resuscitation devices routinely used in the delivery room are capable of tripling the intended TV while providing PPV in a newborn manikin x. Large TV can lead to volutrauma, which is associated with adverse pulmonary outcomes. A study in preterm lambs showed as few as six large tidal volume breaths at birth can lead to acute lung injury and blunt the effect of subsequent surfactant treatment. Ventilation with large breaths may cause gross overexpansion of regions that are forced open, leaving major parts of the lung blocked by fluid and unexpanded, and such regional over distension can be expected to cause epithelial and microvascular injury and pulmonary edema. The resultant pulmonary edema may make the lung more susceptible to further volutrauma during conventional mechanical ventilation. Several animal studies have demonstrated that PPV with TV more than 8 mL/kg causes lung inflammation and lung injury. Additionally, animal and human studies have demonstrated that excessive TV delivery during PPV in the delivery room causes brain inflammation and injury. Likewise, recent meta-analysis data demonstrate infants ventilated using volume targeted ventilation (VTV) modes reduce rates of death or BPD, pneumothoraces, hypocarbia, severe cranial ultrasound pathologies and reduce the duration of ventilation compared with infants ventilated using PLV modes. The risk of lung injury is in all likelihood related to the magnitude of the volutrauma at birth, and therefore ventilation immediately after birth needs to be very gentle.

Without information about TV in the DR and rapidly changing lung compliance, PLV may lead to volutrauma. But no study has specifically evaluated the ability to measure TV provided in intubated infants in the DR or aimed at performing VTV in the DR while assessing its potential role in reducing lung injury.

INNOVATION With recent advances in technology and ability to measure small TV at the endotracheal tube (ET) level with the help of flow sensors, TV can be measured accurately at the ET tube level and volume targeted ventilation (VTV) becomes a possible alternative method of ventilating preterm infants. For the study, infants will have a flow sensor placed in series between the ETT and pressure generating device (T-piece resuscitator, self-inflating bag). The flow sensor will be connected to Respironics NM3 monitor (Philips Healthcare, Eindhoven, Netherlands) to measure the breath to breath TV. The flow sensor adds less than 1 mL of airway dead space volume (Vd) for neonatal sensors (ETT size of 2.5-4 mm). Phase 1 of the study will look into the feasibility of measuring TV in preterm infants. As some of the smallest very low birth weight (VLBW) infants may weight as less as 500gm, goal TV range of 4-6ml/kg will be equal to 2ml-3ml per breath. No study has specifically looked into the ability of measuring such small tidal volume, and hence this feasibility study is of prime importance.

In Phase 2, by using the information of measured TV at the ETT level, the provider can quickly regulate the peak pressure delivered to the infant to achieve a goal TV of 4-6 ml/kg. The provider will be trained to increase or decrease the pressures, by following a strict protocol to ensure the TV remains at goal during neonatal resuscitation. As soon as the infant is stable, the infant will be transitioned to a ventilator with volume targeting capabilities. With stable lung expansion, infants receiving VTV will receive goal TV more consistently, will have reduced incidence of atelectotrauma, volutrauma and overall reduced lung injury with lesser long term pulmonary morbidities.

With the proposed study, in Phase I, the investigators aim to demonstrate that measuring TV in the DR is feasible and is highly variable in the first few hours of life, even with the same peak inspiratory pressures due to rapidly changing pulmonary compliance. A successful Phase I will provide evidence that providing consistent VTV is possible in the DR by adjusting the PiP. In Phase II, the investigators aim to obtain pilot data assessing the feasibility of VTV in the DR, and attempt to understand the pulmonary mechanics and physiology during VTV. A successful pilot study will demonstrate that VTV is feasible; is associated with consistent delivered TV; lower PiP and oxygen needs for the patients; thereby justifying a larger randomized control trial to evaluate the efficacy of VTV in reducing BPD and long term pulmonary morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 32 weeks of gestation
* Infant born at Baystate Medical Center
* Requiring intubation and positive pressure ventilation in the delivery room
* Parental Consent

Exclusion Criteria:

* Maternal prolonged rupture of membrane > 2 weeks duration
* Known congenital or cardiac abnormalities or discovered in the immediate neonatal period.

Ages: 5 Minutes to 60 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Timing of initiation of mechanical ventilation | First 5 mins of life
  The timing of initiation of VTV will be similar to PLV

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Vaidya, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03938532/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03938532/ICF_001.pdf